CLINICAL TRIAL: NCT04723706
Title: Immunological Response to SARS-CoV-2 Vaccine in Stem Cell Transplant and Cellular Therapy Patients
Brief Title: Response to SARS-CoV-2 Vaccine in Stem Cell Transplant and Cellular Therapy Patients
Status: Completed | Type: Observational
Sponsor: Henry Ford Health System (Other)
Responsible Party: Principal Investigator, Shatha Farhan, MD clinical assistant professor, Henry Ford Health System
Other Study IDs: 14632
Record Dates: First submitted 2021-01-20; First posted 2021-01-26 (Actual); Last update posted 2024-04-23 (Actual); Status verified 2024-04

CONDITIONS: Hematologic Disorders and Bone Marrow Failure, Hematopoietic Stem Cell Transplantation (HSCT) or Cellular Therapy (CART)
Keywords: vaccine
MeSH Terms: conditions — Hematologic Diseases; Bone Marrow Failure Disorders

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: COVID-19 serology IgG — patients with SCT or CART who decide to get their vaccines we will measure response by therapy by measuring COVID-19 serology IgG at the following schedule: Baseline +5 days after vaccination; 1 month +/- 10 days (after the first dose), 2 months +/- 10 days (after the 2nd dose), 3 months +/- 10 days, 6 months +/- 10 days and 12 months +/- 10 days

SUMMARY:
For many patients with hematologic disorders and bone marrow failure, hematopoietic stem cell transplantation (HSCT) or cellular therapy (CART) offers a curative treatment option. Patients after SCT or CART have a variable period of immune deficiency in the post-treatment period. The response to vaccination may affect the outcome of the transplant patients. the immunogenicity of vaccines in this immunosuppressed population is uncertain and variable. HSCT and CAR-T recipients are in a COVID-19 high-risk group and conferring immunity by vaccination at the earliest effective timepoint is desirable. At present, the immunogenicity and efficacy of SARS-CoV-2 vaccines in immune-impaired patients including autologous and allogeneic HSCT recipients is unknown. Furthermore, the impact of GvHD and IST on SARS-CoV-2 vaccine immunogenicity is unknown. the investigators aim to evaluate the vaccination response to COVID vaccines after SCT and CART

DETAILED DESCRIPTION:
so for participants with SCT or CART who decide to get their vaccines, the investigators will measure response by therapy by measuring COVID-19 serology IgG at the following schedule: Baseline +5 days after vaccination; 1 month +/- 10 days (after the first dose), 2 months +/- 10 days (after the 2nd dose), 3 months +/- 10 days, 6 months +/- 10 days and 12 months +/- 10 days In addition, also the investigators will collect CD4 and Total IgG which is the standard of care of these patients post SCT and CART

ELIGIBILITY:
Inclusion Criteria:

* any SCT or CART post COVID vaccine

Exclusion Criteria:

* none

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: any SCT or CART post COVID vaccine
Sampling Method: Non-Probability Sample
Enrollment: 33 (Actual)
Dates: Start 2021-03-19 (Actual); Primary Completion 2023-12-02 (Actual); Study Completion 2024-01-02 (Actual)

PRIMARY OUTCOMES:
estimate range for COVID-19 serology IgG in SCT and CART patients post vaccine | up to one year post vaccine

CONTACTS AND LOCATIONS:
Locations (1):
- Henry Ford Health System, Detroit, Michigan, United States

IPD SHARING:
Plan to Share IPD: No